CLINICAL TRIAL: NCT01440725
Title: Multicenter Double Blind, With Evaluator Blinding, Parallel, Randomized Clinical Trial, to Assess the Efficacy of Platelet Rich Plasma for Treatment of Muscle Rupture With Haematoma
Brief Title: Efficacy of Platelet Rich Plasma for Treatment of Muscle Rupture With Haematoma
Acronym: PRP-RICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Terapia Regenerativa Tissular (Other)
Collaborators: Asociacion Colaboracion Cochrane Iberoamericana (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-RICE; ISCIII; Spain (Other Grant/Funding Number: PI080724)
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Muscle Injuries
Keywords: muscle; injuries; platelet-rich plasma; autologous; haematoma
MeSH Terms: conditions — Wounds and Injuries; Hematoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP (Experimental): Administration of 4-8cc of autologous Platelet-rich plasma (PRP)into the muscle wound after the evacuation of the haematoma.
  Interventions: Biological: Autologous Platelet-rich plasma (PRP)
- Evacuation of haematoma (Active Comparator): Evacuation of the hematoma, and simulation of the administration of PRP
  Interventions: Procedure: Evacuation of haematoma

INTERVENTIONS:
Biological: Autologous Platelet-rich plasma (PRP) — 4-8cc, a single dose
  Other Names: Platelet-rich plasma; Growth factors from platelet-rich plasma
  Arms: PRP
Procedure: Evacuation of haematoma — Evacuation of the haematoma, a single procedure
  Other Names: Drainage of haematoma
  Arms: Evacuation of haematoma

SUMMARY:
This is a multicenter, simple blind, masking of outcomes assessors, parallel, randomised clinical trial in patient with muscle rupture and with hematoma production. The main hypothesis is that infiltration in the area of muscle injury in autologous platelet-rich plasma (PRP)improves muscle regeneration and repair by shortening the time to complete recovery.

The main objective is to evaluate the PRP for healing muscular lesions 'tennis leg' type or distal rectus femoral. The secondary objectives are: to evaluate the risk of lesion recurrence; to evaluate the quality of lesion recovery process and evaluate intervention's safety.

Experimental treatment will be the administration of PRP autologous (4-8 cc in a unique dose) by muscular infiltration en the empty space generated after the hematoma evacuation. Control treatment will be hematoma evacuation. Both treatment groups will use compressive bandage and they will recommend rest, extremity elevation, local ice and lately physiotherapy.

Size sample: 76 patients (38 in each group)

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* Lesion with haematoma at the Gastrocnemius muscle or the lower portion of the rectus femoral muscle
* Acceptance to participate at the clinical trial
* Not indicated the surgical treatment of the muscle injury

Exclusion criteria

* Patients who do not meet the inclusion criteria
* History of bleeding disorders
* Inability to follow-up the patient
* The use of corticosteroids, acetylsalicylic acid(Aspirin ®) and nonsteroidal antiinflammatory drugs during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to complete recover of muscular lesions | weekely assessment during 8 weeks
  The complete recovering will be when the patient does his habitual activity.

SECONDARY OUTCOMES:
Percentage of muscular lesion recurrence. | During all study (one year of follow-up)
  Percentage of patients with muscular lesion recurrence.
  Muscular lesion recurrence will be considered if there are symptoms and a lesion gap by ultra sound scan.
Percentage of healing | 8 weeks
  Percentage of patients with the healed lesion
Quality of the regenerated area | at 8 week
  By ultrasonography, the characteristics of the wound will be quantified (size, fibrosis)
Pain | 12 months
  The pain will be measured by a VAS each week, the first 8 weeks of the study and, at 6 and 12 month.
Adverse effects to treatments | 12 months
  Adverse effects will be assessed each week, the first 8 weeks of the study and, at 6 and 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Martínez Zapata, Mª José, Principal Investigator — Centro Cochrane Iberoamericano. Servicio de Epidemiología Clínica y Salud Pública. IIB Sant Pau; Orozco Delclòs, LLuís, Principal Investigator — Institut de Teràpia Regenerativa i Tissular. Centro Médico Teknon. Barcelona
Locations (1):
- Centro Cochrane Iberoamericano, Barcelona, Barcelona, Spain